CLINICAL TRIAL: NCT00716287
Title: Characterisation of Gene Variants in the Angiogenic Pathway
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: MC01/03/07
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Solid Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 1: Anti-angiogenic targeted therapies are used in a wide range of solid tumors including NSCLC, breast cancer, GISTs, CRC, renal cell carcinoma and hepatocellular carcinoma.

SUMMARY:
Anti-angiogenic targeted therapies are used in a wide range of solid tumors including NSCLC, breast cancer, GISTs, CRC, renal cell carcinoma and hepatocellular carcinoma. Somatic mutations in genes related to tumorigenesis have been associated with treatment response whereas germline gene variants have been associated with tumor risk, prognosis and treatment related toxicity.Study objectives are:

1. To characterise the prevalence and clinicopathological associations of germline and somatic variation in genes involved in the angiogenic pathway in healthy donors and unselected cancer patients
2. To examine the association between angiogenic gene variants and outcome in patients receiving anti-angiogenic therapy

DETAILED DESCRIPTION:
Angiogenesis plays a key role in the process of tumour growth and metastases. Anti-angiogenic targeted therapies are currently used in a wide range of solid tumors including lung, breast, colorectal, kidney and liver cancer. Somatic variants in genes related to tumorigenesis have been associated with treatment response, whereas germline gene variants have been associated with tumor risk, prognosis and treatment related toxicity. In this study we propose to (1) To characterise the prevalence and clinicopathological associations of germline and somatic variation in genes involved in the angiogenic pathway in healthy donors and unselected cancer patients (2) to examine the association between angiogenic gene variants and outcome in patients receiving anti-angiogenic therapy. Genes related to angiogenesis to be characterised include those encoding platelet derived growth factor receptors, vascular endothelial growth factors, vascular endothelial growth factor receptors, K-Ras, B-Raf, and c-kit. Results from this study may (1) identify patients who are more likely to respond to anti-angiogenic targeted therapy, thus maximising drug efficacy and (2) to identify further targets for potential anti-angiogenic drug therapies.

ELIGIBILITY:
Inclusion Criteria:

* Anti-angiogenic targeted therapies are used in a wide range of solid tumors including NSCLC, breast cancer, GISTs, CRC, renal cell carcinoma and hepatocellular carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anti-angiogenic targeted therapies are used in a wide range of solid tumors including NSCLC, breast cancer, GISTs, CRC, renal cell carcinoma and hepatocellular carcinoma.
Sampling Method: Non-Probability Sample
Dates: Start 2007-03; Primary Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Andrew Soo, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore